CLINICAL TRIAL: NCT00275561
Title: A Randomized Placebo-controlled Trial of Swallowed Fluticasone in Treatment of Eosinophilic Esophagitis
Brief Title: Topical Steroid Treatment for Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Jeffrey A. Alexander, M.D, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1488-05
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Fluticasone; Dysphagia
MeSH Terms: conditions — Eosinophilic Esophagitis; Deglutition Disorders | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone (Experimental): Aerosolized swallowed fluticasone 880 mcg bid for 6 weeks
  Interventions: Drug: Fluticasone
- Placebo (Placebo Comparator): Placebo inhaler swallowed bid for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone — Aerosolized swallowed fluticasone 880 mg twice a day
  Other Names: Flonase; Veramyst
  Arms: Fluticasone
Drug: Placebo — Placebo inhaler swallowed twice a day for 6 weeks
  Arms: Placebo

SUMMARY:
This was a randomized controlled trial of swallowed fluticasone vs. placebo for eosinophilic esophagitis. Eosinophilic esophagitis is an inflammatory condition in which the wall of the esophagus becomes filled with large numbers of eosinophils, a type of white blood cell. Patients who have this condition have difficulty in swallowing (dysphagia) solid food.

Prior to treatment the patients had biopsies of their esophagus and took questionnaires regarding their symptoms. Treatment was given for 6 weeks, after which biopsies were taken from the esophagus to measure any changes in the tissue from before treatment. The primary endpoint was improvement in dysphagia as measured by the validated Mayo Dysphagia Questionaire. Secondary outcomes included partial symptom response, and histologic (tissue) response to treatment.

DETAILED DESCRIPTION:
This was a double-blind randomized placebo controlled trial to evaluate the effect of aerosolized fluticasone therapy on symptomatic dysphagia and histologic eosinophilia in adults newly diagnosed with eosinophilic esophagitis (EoE). Participants were randomized to receive aerosolized swallowed fluticasone 880 mcg bid or placebo inhaler swallowed bid for 6 weeks.

Four mid esophageal biopsies were obtained from 10 cm above the squamo-columnar junction; then formalin-fixed and stained with hematoxylin and eosin. All esophageal biopsies were read and scored by a single expert gastrointestinal pathologist. The formalin-fixed paraffin-embedded esophageal biopsies were retrieved and underwent standard major basic protein (MBP) immunofluorescence staining. All special stain slides were then read and scored by another pathologist. 24-hour urine was collected for free cortisol by the standard technique. The original endoscopy was performed before the patient was enrolled in the trial by standard clinical technique. The endoscopy post treatment was done in the clinical research unit by the principal investigator.

Patients kept compliance logs that were reviewed at phone interviews at 2 and 4 weeks time and at the end of study evaluation. Ninety percent compliance was required for study inclusion.

At the end of 6 weeks, a 24-hour urine cortisol was done, and patients underwent a repeat endoscopy while still on treatment. Mid-esophageal biopsies were obtained and evaluated for eosinophil density and mast cell degranulation. At this visit the patients returned dysphagia and side effects questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* > 20 eosinophils / hpf on biopsies from mid esophagus (hpf = high-powered field)
* Abnormal dysphagia questionnaire (question 1a "yes", question 1c > "moderate" and question 2 > "less than once a week") on Mayo Dysphagia Questionnaire.

Exclusion Criteria:

* Clinical evidence of infectious process potentially contributing to dysphagia (e.g., candidiasis, cytomegalovirus, herpes)
* Systemic or topical steroid therapy for any reason over the past 3 months
* Previous steroid treatment for Eosinophilic Esophagitis
* Intolerance to steroid therapy in the past
* Other cause of dysphagia identified at endoscopy (e.g., reflux esophagitis, stricture, web, ring, achalasia, esophageal neoplasm)
* Dilatation of esophagus at time of index endoscopy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2005-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Alexander, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] McElhiney J, Lohse MR, Arora AS, Peloquin JM, Geno DM, Kuntz MM, Enders FB, Fredericksen M, Abdalla AA, Khan Y, Talley NJ, Diehl NN, Beebe TJ, Harris AM, Farrugia G, Graner DE, Murray JA, Locke GR 3rd, Grothe RM, Crowell MD, Francis DL, Grudell AM, Dabade T, Ramirez A, Alkhatib M, Alexander JA, Kimber J, Prasad G, Zinsmeister AR, Romero Y. The Mayo Dysphagia Questionnaire-30: documentation of reliability and validity of a tool for interventional trials in adults with esophageal disease. Dysphagia. 2010 Sep;25(3):221-30. doi: 10.1007/s00455-009-9246-8. Epub 2009 Oct 24. PMID 19856027

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with a new diagnosis of eosinophilic esophagitis were recruited at the Mayo Clinic Rochester between 10/2005 and 12/2009.
Period: Overall Study
Arm/Group | Fluticasone | Placebo
Started | 21 | 21
Completed | 19 | 15
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Travel | 1 | 1
Not completed — Scheduling | 1 | 2
Not completed — Family Issues | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age Continuous [Mean (Full Range); unit: years] | 37.5 [19 to 59] | 35 [20 to 57] | 37.5 [19 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 18 | 16 | 34
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42
Food Impaction > 5 minutes [Number; unit: participants] — Food stuck and unable to swallow liquids for >5 minutes
  participants
    Participants with Food Impaction | 16 | 17 | 33
    Participants without Food Impaction | 5 | 4 | 9
Mean Esophageal Eosinophil Count [Mean (Full Range); unit: eosinophils/high powered field] | 40 [8 to 100] | 40 [20 to 80] | 40 [8 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response to Dysphagia
Description: Measured by the Mayo Dysphagia Questionnaire, a validated 28 item instrument; 0=no dysphagia, higher levels indicate greater dysphagia severity. A complete symptom response was defined as an answer of "no" to the question "In the past 2 weeks, have you had trouble swallowing, not associated with other cold symptoms (such as strep throat or mono)?"
Time Frame: 2 weeks
Population: Analysis was run per protocol.
Measure: Number; unit: participants
Arm/Group | Fluticasone | Placebo
Number analyzed (Participants) | 19 | 15
participants | 9 | 6
Statistical Analysis 1: Comparison: Fluticasone vs Placebo; Test type: Superiority or Other; p = 0.74, Fisher Exact

2. Secondary Outcome: Number of Participants With Partial or Complete Response to Dysphagia
Description: Measured by the Mayo Dysphagia Questionnaire, a validated 28 item instrument; 0=no dysphagia, higher levels indicate greater dysphagia severity. A complete symptom response was defined as an answer of "no" to the question "In the past 2 weeks, have you had trouble swallowing, not associated with other cold symptoms (such as strep throat or mono)?" A partial symptom response was defined as an answer of yes to the above question and a decrease in severity of at least 2 levels, or a decrease in frequency of at least 1 level.
Time Frame: 2 weeks
Population: Analysis was run per protocol.
Measure: Number; unit: participants
Arm/Group | Fluticasone | Placebo
Number analyzed (Participants) | 19 | 15
participants | 12 | 7
Statistical Analysis 1: Comparison: Fluticasone vs Placebo; Test type: Superiority or Other; p = 0.49, Fisher Exact

3. Secondary Outcome: Number of Participants With Complete Histologic Response
Description: A complete histologic response was defined as >90% decrease in mean eosinophil count/high powered field
Time Frame: 2 weeks
Population: Analysis was run per protocol.
Measure: Number; unit: participants
Arm/Group | Fluticasone | Placebo
Number analyzed (Participants) | 19 | 15
participants | 13 | 0
Statistical Analysis 1: Comparison: Fluticasone vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Safety was assessed with the side effect questionnaire at weeks 2 and 4 completed by a structured phone interview. The side effect questionnaire had questions on sore throat, hoarseness, white spots in the mouth, irritability, leg swelling, sleep disturbance, appetite change, acne, headache, diarrhea, nausea, and other new symptoms.
Arm/Group | Fluticasone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 7/19 | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone (N=19) | Placebo (N=15)
Sore throat (Gastrointestinal disorders) | 2 (2) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Esophageal candidiasis (Gastrointestinal disorders) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
The relatively small sample size; unexpected high dropout rate in the placebo group; study commenced before the consensus definition of EoE advising exclusion of gastroesophageal reflux disease (GERD) was established.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes